CLINICAL TRIAL: NCT00874796
Title: A Phase 2b, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of GS 9450 in Adults With Chronic Hepatitis C Virus Infection (GS-US-227-0106)
Brief Title: Efficacy and Safety Study of GS-9450 Treatment for 6 Months in Patients With Chronic Hepatitis C Virus Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Reports of significant laboratory abnormalities and adverse events in a number of clinical study participants.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-227-0106
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: HCV Infection
Keywords: apoptosis; liver inflammation; hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GS-9450 10 mg/day (Experimental): GS-9450 taken as one 10 mg capsule by mouth once daily
  Interventions: Drug: GS-9450
- GS-9450 40 mg/day (Experimental): GS-9450 taken as one 40 mg capsule by mouth once daily
  Interventions: Drug: GS-9450
- Placebo (Placebo Comparator): Placebo taken as one placebo capsule by mouth once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-9450 — Taken as one capsule by mouth once daily
  Arms: GS-9450 10 mg/day; GS-9450 40 mg/day
Drug: Placebo — Taken as one placebo capsule (matching in appearance to GS-9450 capsules) by mouth once daily
  Arms: Placebo

SUMMARY:
This is a Phase 2b, randomized, double-blind, parallel-group, placebo-controlled, multicenter study investigating the safety, tolerability and efficacy of two oral doses of GS-9450 in adults with chronic Hepatitis C Virus (HCV). Approximately 240 subjects 18-65 years of age who meet study entry criteria will be randomized (in other words, selected at random, like flipping a coin) to one of three treatment groups (80 subjects per treatment group) as follows:GS-9450 10 mg once daily,GS-9450 40 mg once daily, or matching placebo once daily.

Following randomization, subjects will return within seven business days for a Baseline (Day 1) visit, at which time study medication will be dispensed and subjects will enter a 26 week treatment phase. During the treatment phase, subjects will receive study drug once daily for 24 weeks and then taper off of study drug over the following 2 weeks by receiving study drug once every other day for one week and then every 3 days for one week. Following completion of the treatment phase, subjects will enter a 4-week off-treatment follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, ages 18-65
* Chronic HCV infection, defined as having documented HCV infection (antibody or RNA positivity) at least 6 months prior to Baseline (Day 1) with HCV viremia at screening
* Screening Knodell necroinflammatory score >= 3 based on liver biopsy evaluation (as determined by local pathologist) conducted anytime during the 45-day screening period
* ALT > the upper limit of the normal range (ULN) but < 10 X ULN at the screening visit
* Previously failed pegylated interferon-based HCV therapy in combination with ribavirin therapy, or is unable to tolerate or has contraindications to receiving interferon or ribavirin therapy
* BMI between 19 and 36 kg/m2 (inclusive)
* Creatinine clearance >= 70 mL/min
* absolute neutrophil count >= 1000/mm3
* Hemoglobin > 10 g/dL
* Have no clinical or laboratory evidence of hepatic decompensation

Exclusion Criteria:

* Decompensated liver disease
* Child-Pugh grade B or C cirrhosis
* Evidence of hepatocellular carcinoma
* Positive urine drug screen for cocaine or amphetamines
* Infection with HCV genotype 3
* Co-infection with hepatitis B virus or human immunodeficiency virus
* Pancreatitis
* Recent significant infection or symptoms of infection
* Autoimmune disorders
* Any history of seizure
* Is a public transportation operator (pilot of airplane or ship; air traffic controller; bus, train or subway driver) or operates heavy construction machinery
* Transplantation
* History of malignancy
* Current excessive alcohol ingestion, averaging > 3 drinks/day for females and > 4 drinks/day for males
* History of or current binge drinking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Histologic response, defined as a >= 2-point decrease in Knodell necroinflammatory score with no concurrent worsening in the Knodell fibrosis score, at Week 24 . | Week 24 on-treatment

SECONDARY OUTCOMES:
Change (absolute, percent) from baseline in the Knodell necroinflammatory score | Baseline to Week 24
Change (absolute, percent) from pretreatment in alanine aminotransferase (ALT) levels | Baseline to Week 24
Percentage of Participants Who Experienced Adverse Events (AEs) and Graded Laboratory Abnormalities | Up to 24 weeks plus 30 days following the last dose of study drug
Change (absolute, percent) from baseline in cytokeratin-18 caspase cleavage fragment levels | Baseline to Week 24
Change from baseline in hepatic collagen staining area as measured by morphometry of liver biopsy specimens | Baseline to Week 24
Change from baseline in the percent of apoptotic cells | Baseline to Week 24
  Change from baseline in the percent of apoptotic cells (transferase deoxyuridine triphosphate [dUTP] nick end labeling [TUNEL] positive) as measured by TUNEL staining of liver biopsy specimens
Change from baseline in percent of anti-M30 monoclonal antibody-positive hepatocytes | Baseline to Week 24
  Change from baseline in percent of anti-M30 monoclonal antibody-positive hepatocytes (for cytokeratin-18 neoantigen expression) as measured by immunohistochemical staining of liver biopsy specimens
Change From Baseline in HCV RNA | Baseline to to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Ken Hirsch, MD, Study Director — Gilead Sciences
Locations (73):
- United States (51):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Beverly Hills, California
  - Cypress, California
  - La Jolla, California
  - Mission Hills, California
  - Palm Springs, California
  - Pasadena, California
  - San Clemente, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - Hialeah, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Novi, Michigan
  - Saint Louis, Michigan
  - Plymouth, Minnesota
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Hillsborough, New Jersey
  - Morristown, New Jersey
  - Santa Fe, New Mexico
  - Johnson City, New York
  - New York, New York
  - Plainview, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Canada (3):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - London, Ontario
- Germany (8):
  - Berlin
  - Bonn
  - Cologne
  - Essen
  - Frankfurt am Main
  - Hamburg
  - Hanover
  - Mainz
- Poland (5):
  - Bialystok
  - Bydgoszcz
  - Chorzów
  - Kielce
  - Wroclaw
- Puerto Rico (2):
  - San Juan
  - Santurce
- United Kingdom (4):
  - Brighton
  - London
  - Nottingham
  - Sheffield